CLINICAL TRIAL: NCT03427112
Title: Clinical Validation of the Xin1 Humerus System
Brief Title: Assessment of the Surgical Handling and Performance of the X-ray-based Tracking and Navigation System "Xin1 Humerus System" Evaluated From 10 Proximal Humerus Plate Fixations
Status: Completed | Type: Observational
Sponsor: AO Research Institute Davos (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Xin1Humerus; 80M0661 (Other: FAGG (Federal agency for medicines and health products, Brussels, Belgium))
Record Dates: First submitted 2018-01-18; First posted 2018-02-09 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Xin1 Humerus System — Retrospective assessment of the surgical handling and performance of the X-ray-based tracking and navigation system "Xin1 Humerus system" evaluated from 10 proximal humerus plate fixations

SUMMARY:
Xin1 Humerus system is an X-ray-based tracking and navigation system designed to calculate the plate position and all required proximal screw lengths for proximal humerus plate fixation. The aim is to validate the system performance in a clinical context and test the surgical handling of the Xin1 marker in a hospital environment. 10 adults having sustained a proximal humerus fracture and are indicated for plate fixation osteosynthesis will be provided intraoperatively with the Xin1 marker. The system performance is evaluated retrospectively by post-processing the intraoperative X-ray images after surgery

DETAILED DESCRIPTION:
Treatment of fragility fractures at the proximal Humerus still remains a major challenge in trauma surgery. Several factors such as highly compromised bone mass, complex loading conditions, multi-fragment fractures, absent bony support and limited surgical access render the fixation particularly complex. Especially in elderly osteoporotic patients, implant position and fixation plays a key role for a successful outcome. Nowadays, complication rates of plate and screw fixation systems in the proximal Humerus region under complex fracture patterns are reported to range between 28% and 79%. A significant portion of these cases can be attributed to implant mal-placement. Particularly, when screws are too short and the subchondral bone stock is missed out, screw anchorage is significantly compromised. On the other hand, if screws are too long they might penetrate into the joint with devastating consequences. Adequate selection of screw length is hence of utmost importance. However, the particular anatomical situation challenges the determination procedure which results in prolonged operational time and increased X-ray exposure. New strategies are needed to simply, reliably and accurately fix proximal humeral fractures with plate-screw constructs. Xin1 is an X-ray-based tracking and navigation system designed to simplify a variety of surgical applications. For the Humerus application the position in space of the proximal Humerus plate is calculated in such manner, which then can be related to the position of the humeral head as derived from an image pair. All required proximal screw lengths are determined from these two radiographs. From ex-vivo evaluation the Xin1 Humerus System has proven its value in terms of accuracy increase as well as time and X-ray reduction. A clear potential for improving clinical practice is therefore apparent. The consequent next step is a first clinical phase verifying the basic function of the Xin1 system in a clinical context and investigating the surgical handling in a hospital environment.

This clinical trial aims to

1. validate the Xin1 Humerus system performance in a clinical context.
2. test the surgical handling of the Xin1 marker in a hospital environment.

There is no additional time effort required from the patient. All capacitated adults having sustained a proximal humerus fracture indicated for plate fixation osteosynthesis can be included in the study. The study is limited to 10 patients and 1 year. To minimize the patient risk it is suggested in this first study phase to entirely eliminate the system feedback to the surgeon during surgery. The system performance is evaluated retrospectively by post-processing X-ray images after surgery. The Xin1 system used during surgery is thereby reduced to the Xin1 marker clip (REF 100838-00) only.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of proximal humerus fracture
* Indicated for plate fixation osteosynthesis
* Informed consent obtained

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with proximal humerus fracture which are transferred to the Dpt. Traumatologie, ZU Leuven, will be recruited during diagnosis and indication.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Influence of plate fixation on the determined screw lengths derived from the Xin1 Humerus System | during surgery
  Xin1 Humerus System:
  * Screw lengths determined after fracture reduction and temporary fixation
  * Screw lengths determined after final plate fixation

SECONDARY OUTCOMES:
Treatment information | during surgery
  * Fracture classification according to AO
  * Anatomical side of the fracture
  * Actual screw lengths of the implanted screws
  * Cumulative fluoro time
  * Cumulative area dose product
  * Brand and Model of used C-arm
Patient information | Preoperative
  * Gender
  * Age
System information | during surgery
  • Accuracy estimation of the Xin1 Humerus System in terms of screw length prediction in the humeral head.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan Nijs, Prof., Principal Investigator — UZ Leuven campus Gasthuisberg
Locations (1):
- UZ Leuven campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voigt C, Woltmann A, Partenheimer A, Lill H. [Management of complications after angularly stable locking proximal humerus plate fixation]. Chirurg. 2007 Jan;78(1):40-6. doi: 10.1007/s00104-006-1241-0. German. PMID 16998660
- [Background] Solberg BD, Moon CN, Franco DP, Paiement GD. Locked plating of 3- and 4-part proximal humerus fractures in older patients: the effect of initial fracture pattern on outcome. J Orthop Trauma. 2009 Feb;23(2):113-9. doi: 10.1097/BOT.0b013e31819344bf. PMID 19169103